CLINICAL TRIAL: NCT04390334
Title: Single-center, Randomized, Open-label Study to Investigate the Effect of Single-dose Famotidine and Multiple-dose Efavirenz on the Pharmacokinetics of Daridorexant in Healthy Male Subjects
Brief Title: A Study in Healthy Male Subjects to Investigate the Effect of Famotidine and Efavirenz on the Way the Body Takes up, Distributes, and Gets Rid of Daridorexant.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ID-078-120; 2020-000653-27 (EudraCT Number)
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Healthy
MeSH Terms: interventions — daridorexant; Famotidine; efavirenz

STUDY DESIGN:
Intervention Model Description: 4 treatment arms in 2 sequences, ABCD or BACD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A: Daridorexant (Experimental): Single dose of 50 mg daridorexant
  Interventions: Drug: Daridorexant
- Treatment B: Famotidine & daridorexant (Experimental): Single dose of 40 mg famotidine followed 3 h later by a single dose of 50 mg daridorexant
  Interventions: Drug: Daridorexant; Drug: Famotidine
- Treatment C: Efavirenz (Experimental): 600 mg efavirenz once daily in the evening from Day 5 to Day 14
  Interventions: Drug: Efavirenz
- Treatment D: Daridorexant & efavirenz (Experimental): Single dose of 50 mg daridorexant in the morning of Day 15 followed by a single dose of 600 mg efavirenz in the evening of Days 15 and 16
  Interventions: Drug: Daridorexant; Drug: Efavirenz

INTERVENTIONS:
Drug: Daridorexant — Daridorexant will be administered orally as 1 film-coated tablet of 50 mg strength to be taken in the morning under fasted conditions.
  Arms: Treatment A: Daridorexant; Treatment B: Famotidine & daridorexant; Treatment D: Daridorexant & efavirenz
Drug: Famotidine — Famotidine will be administered orally as 1 film-coated tablet of 40 mg strength to be taken in the morning under fasted conditions.
  Arms: Treatment B: Famotidine & daridorexant
Drug: Efavirenz — Efavirenz will be administered orally as 1 film-coated tablet of 600 mg strength o.d. in the evening.
  Arms: Treatment C: Efavirenz; Treatment D: Daridorexant & efavirenz

SUMMARY:
A study in healthy male subjects to investigate the effect of famotidine and efavirenz on the way the body takes up, distributes, and gets rid of daridorexant.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Healthy male subjects aged between 18 and 45 years (inclusive) at Screening.

Exclusion Criteria:

* Clinically relevant findings on the physical examination at Screening.
* Clinically relevant abnormalities on 12-lead ECG, measured after at least 5 min in a supine position at Screening.
* Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry) at Screening and on Day -1.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment(s) (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Moderate or severe renal insufficiency (creatinine clearance < 60 mL/min calculated with the Cockcroft Gault formula) at Screening.
* Total bilirubin > 1.5 x Upper Limit of Normal at Screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
PK parameter of daridorexant: Maximum plasma concentration (Cmax) | Various time points during Treatment A through D (Total duration: up to 3 weeks).
PK parameter of daridorexant: Time to reach Cmax (tmax) | Various time points during Treatment A through D (Total duration: up to 3 weeks).
PK parameter of daridorexant: AUC from zero to infinity (AUC0-inf) | Various time points during Treatment A through D (Total duration: up to 3 weeks).
PK parameter of daridorexant: AUC from zero to 48 hours (AUC0-48) | Various time points during Treatment A through D (Total duration: up to 3 weeks).
PK parameter of daridorexant: Terminal elimination half-life (t½) | Various time points during Treatment A through D (Total duration: up to 3 weeks).

SECONDARY OUTCOMES:
Treatment-emergent (S)AEs | Up to EOP for each of the Periods 1 to 3 and up to EOS for Period 4 (Total duration: up to 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Study Director, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No